CLINICAL TRIAL: NCT00573430
Title: A 28-week, Randomised, Open-label, Parallel-Group, Multi-Center Study To Find the Effective Dose of Candesartan Cilexetil (Atacand) for Renoprotection in Korean Hypertensive Patients With Non-diabetic Nephropathy
Brief Title: ARIA (Atacand Renoprotection In NephropAthy Pt.)
Acronym: PCR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2452L00015
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Non-diabetic Nephropathy With Hypertension
Keywords: Candesartan Cilexetil; Non-diabetic Nephropathy; hypertension; urine protein creatinine ratio
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Candesartan Cilexetil
  Interventions: Drug: Candesartan Cilexetil
- 2 (Experimental): Candesartan Cilexetil
  Interventions: Drug: Candesartan Cilexetil
- 3 (Experimental): Candesartan Cilexetil
  Interventions: Drug: Candesartan Cilexetil 32mg

INTERVENTIONS:
Drug: Candesartan Cilexetil — 8 mg oral once daily dose
  Other Names: Atacand
  Arms: 1
Drug: Candesartan Cilexetil — 16 mg oral once daily dose
  Other Names: Atacand
  Arms: 2
Drug: Candesartan Cilexetil 32mg — 32 mg oral once daily dose
  Other Names: Atacand
  Arms: 3

SUMMARY:
To determine the effective dose of candesartan cilexetil for reduction of urinary protein excretion in hypertensive patients with non-diabetic chronic kidney disease with baseline urinary protein/creatinine ratio between 500mg/g and 5000mg/g, by assessing the change in urinary protein/creatinine ratio from baseline to the end of 28-week treatment

ELIGIBILITY:
Inclusion Criteria:

* hypertension; a)135mmHg < Systolic Blood Pressure <180mmHg and/or 85 mmHg < Diastolic Blood Pressure <100 mmHg. or b) The subject has been treated with antihypertensive medication
* proteinuria (urinary protein/creatinine ratio between 500 mg/g and 5000 mg/g)

Exclusion Criteria:

* Current serum-creatinine > 265 mmol/L (>3 mg/dL).
* Current serum-potassium > 5.5 mmol/L
* Known hypersensitivity to angiotensin (AT)1-receptor blocker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Da Suk Han, Principal Investigator — Severance Hospital
Locations (1):
- Research Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 155 enrolled, 27 screening failure, 128 randomized. Eligibility criteria not fulfilled meant subjects who were not fulfilled at Visit 1 or Enrolment, but screening failure subjects were who fulfilled at Visit 1, but not at Visit 2 after screening period.
Pre-assignment Details: Total 128 patient enrolled, but among of them, 9 subjects excluded from analysis because of Withdrawal by Subject, Protocol violation, Eligibility criteria not fullfiled. You can see these number in above table. This analysis was conducted based on Intend to treat. Therefore, total analyzed number is 119, and 39, 44, 36 per arm respectively.
Groups:
- Candesartan 8 mg: Candesartan 8 mg oral once daily dose
- Candesartan 16mg: Candesartan 16mg oral once daily dose
- Candesartan 32mg: Candesartan 32mg oral once daily dose
Period: Overall Study
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg
Started | 40 (randomized) | 45 (randomized) | 43 (randomized)
Completed | 39 | 40 | 33
Not Completed | 1 | 5 | 10
Not completed — Incorrect enrollment of randomization | 0 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg | Total
Number analyzed (Participants) | 40 | 45 | 43 | 128
Age Continuous [Mean (Standard Deviation); unit: years]
  19 to 70 | 45.70 (11) | 46.80 (16) | 49.50 (11) | 47.3 (13.4)
Gender [Number; unit: Participants] — Analyzed efficacy data and demography data based on Intended to Treat (ITT) set. The discrepancy of "Total" and "Started Period 1" is who is excluded to the ITT set.
  Participants
    Female | 20 | 16 | 17 | 53
    Male | 19 | 28 | 19 | 66

OUTCOME MEASURES:

1. Primary Outcome: The Change in Urinary Protein/Creatinine Ratio From Baseline to 28 Weeks
Description: Decrease of urinary protein/creatinine ratio means improvement of renal disease.
Time Frame: baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg
Number analyzed (Participants) | 39 | 44 | 36
mg/g | 794.0 (1,070.10) | 639.9 (863.30) | 819.0 (823.60)

2. Secondary Outcome: Change of Systolic and Diastolic Blood Pressure From Baseline
Time Frame: baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg
Number analyzed (Participants) | 39 | 44 | 36
mmHg
  Systolic | -11.70 (14.90) | -13.30 (14.90) | -16.10 (17.30)
  Diastolic | -8.90 (13.30) | -8.00 (13.30) | -13.00 (14.70)

3. Secondary Outcome: Inflammatory Marker (Hs-C-peptide Reactive Protein)
Description: To evaluate how to reduce and relate with cardiovascular risk
Time Frame: baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg
Number analyzed (Participants) | 38 | 41 | 35
mg/dL | 0.01 (0.12) | -0.17 (1.86) | -0.01 (0.38)

4. Secondary Outcome: Estimated GFR Predicted From the Modification of Diet in Renal Disease (MDRD) Equation
Description: GFR (mL/min/1.73 m2) = 186 x (Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if African-American) (conventional units)
Time Frame: 28 weeks
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m2
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg
Number analyzed (Participants) | 39 | 44 | 36
mL/min/1.73 m2 | 1.28 (8.45) | 1.20 (9.31) | 0.56 (8.92)

5. Secondary Outcome: Treatment-emergent Adverse Events
Description: Prevalence of adverse events after treatment regardless causality. An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition from the signing of the informed consent, whether or not considered causally related to the product.
Time Frame: Baseline to 28 weeks
Measure: Number; unit: Participants
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg
Number analyzed (Participants) | 40 | 43 | 47
Participants | 28 | 27 | 25

ADVERSE EVENTS:
Arm/Group | Candesartan 8 mg | Candesartan 16mg | Candesartan 32mg
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/45 | 1/43
Other Adverse Events (participants affected / at risk) | 11/40 | 6/45 | 9/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan 8 mg (N=40) | Candesartan 16mg (N=45) | Candesartan 32mg (N=43)
dizziness (Nervous system disorders) | 0 | 1 | 0
Acute leukaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pnuemonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan 8 mg (N=40) | Candesartan 16mg (N=45) | Candesartan 32mg (N=43)
Nasopharyngitis (Infections and infestations) | 4 | 2 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 3
Headache (Nervous system disorders) | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less